CLINICAL TRIAL: NCT04413084
Title: Effects of Vestibular Rehabilitation for Dizziness in Hearing Impaired Children.
Brief Title: Vestibular Rehabilitation for Dizziness in Hearing Impaired Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00653 Poshmal butt
Record Dates: First submitted 2020-04-14; First posted 2020-06-02 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: HEARING IMPAIRED CHILDREN
Keywords: Dizziness; Hearing Impaired children; Vestibular rehabilitation
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaze stability exercises (Experimental): Group I will receive Gaze stability exercises.
  Interventions: Other: Gaze stability exercises
- Brandt-Daroff Exercises (Experimental): Group II will receive Brandt-Daroff Exercises.
  Interventions: Other: Brandt-Daroff Exercises

INTERVENTIONS:
Other: Gaze stability exercises — Business card will be placed at eye level. Begin with simpler exercises and progress toward harder one.
  Arms: Gaze stability exercises
Other: Brandt-Daroff Exercises — Brandt-Daroff Exercises
  1. Start sitting upright on the edge of the bed.
  2. Turn your head 45 degrees to the left, or as far as is comfortable.
  3. Lie down on your right side.
  4. Remain in this position for 30 seconds or until any dizziness has subsided.
  5. Sit up and turn head back to center.
  6. Turn your head 45 degrees to the right, or as far as is comfortable.
  7. Lie down on your left side.
  8. Remain in this position for 30 seconds or until any dizziness has subsided.
  9. Sit up and turn head back to center.
  Arms: Brandt-Daroff Exercises

SUMMARY:
There is a need to manage dizziness in vestibular dysfunction patients with the vestibular rehabilitation to improve the life style of these patients. Vestibular rehabilitation exercises are beneficial for the vestibular dysfunction patients because they decrease dizziness and visual symptoms, increase walking and balance functions and with this the general activity level also increases. In my study my goal is to apply two different vestibular exercise and check their effects on dizziness in hearing impaired children's.

DETAILED DESCRIPTION:
Dizziness is not a disease it is one of the most common symptoms of vestibular dysfunction. There are mainly two types of vestibular dysfunction central and peripheral vestibular dysfunction. Signs of vestibular dysfunction are vertigo, nystagmus, visual instability on head movement, spinning, double vision, May or may not have hearing loss or tinnitus. Due to these problem the patient feel difficulty in movements and in other activities, asymmetrical posture in sitting or standing. patients who experience dizziness report a significant disability that reduces their quality of life.

Vestibular system is consist of two parts central vestibular system and peripheral vestibular system. Peripheral part is consist of three semi-circular canals and otolith organs. The three semi-circular canals horizontal, posterior and anterior respond to angular acceleration and are right angle to one another. Semi-circular canals are filled with endolymph. Which move freely within each canal in response to the direction of the angular head rotation. The saccule and utricle make up the otolith organ which respond to the linear acceleration and the static head tilt. Three main functions of the peripheral vestibular system is stabilize visual images during head movement, maintain postural stability during head movement and providing information about the environment. In the central vestibular system brainstem processes provide primary control of many vestibular reflex. Connection with the thalamus, vestibular cortex and reticular system enable the vestibular system to aware of arousal and conscious awareness of the body and discrimination between the self and environment.

In children, vestibular function plays an important role in postural and gross motor development control. Children with congenitally profound hearing loss suffer vestibular dysfunction in both ears, and loss of postural control. Maintaining and development of postural stability is a multisystem process it does not only depend on vestibular input. Maturational changes in proprioceptive and visual, central nervous system processing, and coordination of motor output are responsible for the changes in postural skills observed through adolescence. Infants and young children are dependent on the visual system to maintain balance. As they grow older, begin to use somatosensory and vestibular information properly. Between the 3 sensory inputs in children, the vestibular system seems to be the slightest effective in postural control.

Children with early sensorineural hearing loss and bilateral vestibular dysfunction present with delayed gross motor development. These children stand and walk later than their peers. Difficulties in maintaining balance can lead to challenges in normal childhood activities e.g. riding a bicycle or hopping. Reduced ability to participate in normal play with other children may result in social isolation. In hearing impaired children vestibular dysfunction is common. It was mentioned in a study held in 2013 that 88% of hearing impaired children suffer from vestibular dysfunction. This could mainly be due to hearing and vestibular impulses pass via the vestibule-cochlear nerve. Another study in 2018, found that vestibular dysfunction to be around 50% in hearing impaired children.

Gaze stability and Brandt-Daroff exercises are two different type of exercises which are used for rehabilitation of dizziness in hearing impaired patients. A type of habituation exercise is Brandt- Daroff exercises which are easy to perform. Brandt- Daroff exercises cause the debris to get dislodged from the cupula of the posterior semi-circular canal and will no longer effect cupula during the head movements. Bandt-Daroff exercises are performed with quick head rotations while watching a visual target and sustaining focus on the visual target during head movements. Gaze stability exercises designed to improve the gaze stability. These exercises require the individual to fixate on a visual target during horizontal or vertical head movement.

ELIGIBILITY:
Inclusion Criteria:

* Children with hearing impairment of both genders, those diagnosed with vestibular dysfunction by ear nose and throat specialist.
* Bilateral hearing loss
* Mild to moderate hearing loss
* Age between 8 to 17 years.
* Any test of the following four tests positive (Dix Hall Pike test, Supine Roll's test, Fukuda Stepping Test and Sharpened Romberg's test) were included in the study

Exclusion Criteria:

* Children receiving some other form of treatment for vestibular dysfunction.
* Suffering from other systemic disorders.
* Musculoskeletal disorders like fractures, strains, sprains leading to imbalance, central or peripheral neurologic diseases leading to disturbed balance.
* Those who were handicapped were excluded from the study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Dix Hall Pike Test | Change from Baseline dizziness and balance to 2 Weeks
  The Dix hall pike test is a diagnostic procedure. When performing the test, patients are lowered quickly to supine position with 30 degrees neck extension below horizontal by the clinician. Positive test is reported when the patients report of a production of vertigo and observation of nystagmus.
Fukuda Step Test | Change from Baseline dizziness to 2 Week
  A vestibulospinal test, fukuda test is used to measure asymmetrical labyrinthine function. One's ability to step in place with eyes closed without turning depends on normal vestibulospinal and proprioceptive function.
Motion Sensitivity Quotient | Change from Baseline dizziness to 2 Week
  Motion Sensitivity Quotient: is a clinical protocol designed to measure motion provoked dizziness during a series of quick changes to head or body position. Test is used as a guide for exercise developing for the patients problems with the motion provoked dizziness, also for the effectiveness of rehabilitation therapy

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | Change from Baseline dizziness to 2 Week
  Dizziness Handicap Inventory: is a self-assessment inventory designed to evaluate the effect of dizziness and unsteadiness. Graded on a scale of 0-100, higher score shows greater perception of handicap due to dizziness
Sharpened Romberg's Test | Change from Baseline balance to 2 Week
  : is an appropriate tool to diagnose gait disturbance caused by abnormal proprioception involving information about the joints. Patients is ask to stand quietly with eyes closed. Patients tries to maintain his balance. The score is counted by the time the patients is able to stand with the eyes closed. A positive sign is noted when a sway is noted with the closed eyes.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- . National Special Education Center Muzaffarabad department of social welfare & women development., Muzaffarabad, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khandare S, Gonsalves N, Palekar DT, Rathi DM, Desai R, Deshmukh MJIJoCRiLS. Efficacy of two different vestibular rehabilitation approaches for dizziness in vestibular dysfunction in hearing impaired children". 2018;7(05):1985-8.
- [Background] Hsiao CJ, Cherry DK, Beatty PC, Rechtsteiner EA. National Ambulatory Medical Care Survey: 2007 summary. Natl Health Stat Report. 2010 Nov 3;(27):1-32. PMID 21089986
- [Background] Lakhani H, Saxena PP, Shethia UJp. Effectiveness of Brandt-daroff exercises on hearing impaired children: A Comparative Study.2:100.
- [Background] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090
- [Background] Suarez H, Angeli S, Suarez A, Rosales B, Carrera X, Alonso R. Balance sensory organization in children with profound hearing loss and cochlear implants. Int J Pediatr Otorhinolaryngol. 2007 Apr;71(4):629-37. doi: 10.1016/j.ijporl.2006.12.014. Epub 2007 Feb 2. PMID 17275927